CLINICAL TRIAL: NCT05961865
Title: Change in Inflammatory State in Patients Undergoing Transcatheter Ablation of Atrial Fibrillation
Acronym: POLICARDIOFA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Stefano Carugo, Director of the Department of Cardio-Thoracic-Vascular Diseases, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 6672
Record Dates: First submitted 2023-07-09; First posted 2023-07-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Marker of Inflammation; Inflammation; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Inflammation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood aliquot will be analyzed for the evaluation of markers of atrial inflammation and fibrosis identified so far in the literature, such as Interleukin 6, N-terminal propeptide of procollagen type 1 (P1NP), chitinase-3-like protein 1 (YKL-40), tumor necrosis factor (TNF-alpha) , GlycA, proprotein convertase subtilisin/kexin type 9 and omega-3 fatty acids.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Markers of inflammation and fibrosis — Will be analyzed the following inflammation markers:
  Interleukin 6, N-terminal propeptide of type 1 procollagen (P1NP), chitinase-3-like protein 1 (YKL-40), tumor necrosis factor (TNF-alpha), GlycA, proprotein convertase subtilisin/kexin type 9 and omega-3 fatty acids.

SUMMARY:
It is a non-pharmacological (biological), spontaneous observational study. The main objective is to evaluate the correlation between inflammation markers and local adiposity, clinical risk factors and their possible variation following an AF ablation procedure

DETAILED DESCRIPTION:
The study includes the execution of a sample for each time point for the evaluation of inflammation and fibrosis markers identified so far in the literature, such as Interleukin 6, N-terminal propeptide of procollagen type 1 (P1NP), chitinase-3-like protein 1 (YKL-40), tumor necrosis factor (TNF-alpha), GlycA, proprotein convertase subtilisin/kexin type 9 and omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent AF;
* Patients undergoing ESC/ERAH(European Society of Cardiology/European Heart Rhythm Association) approved catheter ablation procedures;
* Aged between 18 and 85 years;
* Ability to provide informed consent for study participation.

Exclusion Criteria:

* Age > 85 years or < 18 years;
* Presence of left auricular thrombosis on pre-procedural transesophageal echocardiogram;
* NYHA functional class IV;
* Left ventricular ejection fraction <30%;
* Myocardial infarction or unstable angina or recent coronary artery bypass graft (<6 months);
* Significant co-morbidity, such as cancer, severe renal failure requiring dialysis, severe obstructive pulmonary disease, cirrhosis, with a life expectancy of less than 12 months;
* Presence of contraindications to the procedure;
* Inability to provide informed consent for study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Paroxysmal or Persistent Atrial Fibrillation
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of subjects with AF undergoing ablation who have a reduction of inflammatory burden following treatment. | One year
  Outcome measured through biochemical analyzes conducted on the patient: interleukin 6 (pg/ml), procollagen type 1 N-terminal propeptide (µg/l), chitinase-3-like protein 1(ng/ml), tumor necrosis factor -TNF-alpha - (pg/ml), GlycA (mmol/mol).

SECONDARY OUTCOMES:
Prevalence of subjects with AF undergoing ablation who show improvement in clinical terms and in the arrhythmia recurrence rate. | One year
  Identify how many AF patients undergoing ablation have a reduction in related symptoms such as shortness of breath, feeling tired and weakness. The patient will answer an EQ-5D-5L questionnaire for symptom assessment
Relationship between the degree of inflammation and atrial fibrosis and the degree of atrial fibrosis detected by electroanatomical mapping. | One year
  Relationship between the degree of inflammation and atrial fibrosis detected through biochemical analyzes conducted on the patient: interleukin 6 (pg/ml), procollagen type 1 N-terminal propeptide (µg/l), chitinase-3-like protein 1(ng/ml), tumor necrosis factor -TNF-alpha - (pg/ml), GlycA (mmol/mol) and the degree of atrial fibrosis detected on mapping electroanatomical (voltage map)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Carugo, MD, Principal Investigator — IRCCS Fondazione Cà Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No